CLINICAL TRIAL: NCT01398826
Title: A Pilot Study Assessing the Glycemic Response and Its Relationship to Performance During Road Cycling in Elite Athletes With Type 1 Diabetes and Non-Diabetic Controls
Brief Title: Glycemic Response to Road Cycling in Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Team Type 1, Inc. (Other)
Responsible Party: Juan Pablo Frias, MD, TeamType 1
Other Study IDs: TT1-001
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Exercise; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the glycemic response to cycling road races (using continuous glucose monitoring ) in elite athletes with type 1 diabetes and non-diabetic controls. The investigators will also assess the relationship between power/work during cycling (using a power meter) and the subject's glucose profile.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* A1C ≤8.0% if diagnosed with type 1 DM

Exclusion Criteria:

* If diagnosed with type 1 diabetes, has had recurrent severe hypoglycemia (greater than 2 episodes in previous 6 months requiring assistance by a third party)
* Has any medical condition or medical history that may affect successful completion of the study and/or personal well-being (as assessed by the PI)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professional cyclists on TeamType 1 cycling teams
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Frias, MD, Principal Investigator — Team Type 1, Inc.